CLINICAL TRIAL: NCT00232388
Title: Phase 1 Study of PICP Serum Marker of Myocardial Fibrosis and Diastolic Function in Patients With Systolic Dysfunction
Brief Title: Association of PICP Serum Marker in Patients With LVSD
Status: Terminated | Type: Observational
Why Stopped: PI left institution; Data collected from 45 participants, but no results are available.
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Chanwith Roongsritong, MD
Other Study IDs: L06-006
Record Dates: First submitted 2005-10-03; First posted 2005-10-04 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Systolic Dysfunction
Keywords: Ejection Fraction <35%
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Biospecimen Retention: None Retained — PLEASE NOTE THAT THE INVESTIGATOR LEFT THE INSTITUION WITHOUT PROVIDING ANY INFORMATION REGARDING THIS PROJECT. NO FORWARDING INFORMATION IS AVAILABLE FROM THE INVESTIGATOR.
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood draw

SUMMARY:
The purpose of this study is to determine if the carboxy-terminal of procollagen type I (PICP) can be a useful marker of different degrees of myocardial fibrosis.

DETAILED DESCRIPTION:
Abnormality of diastolic function, particularly a more advanced form known as restrictive tilling pattern, has been correlated with worse outcome in patients with systolic dysfunction associated with chronic heart failure or following an acute myocardial infarction. Recently, the severity of diastolic dysfunction has also been shown to predict the response to cardiac synchronization therapy for refractory heart failure due to systolic dysfunction.

Varying degree of diastolic dysfunction has been reported among patients with comparable severity of systolic dysfunction. The underlying mechanisms responsible for the observed discordance between systolic and diastolic dysfunction in these patients remains incompletely understood.

The carboxy-terminal of procollagen type I (PICP), a peptide that is cleaved from procollagen type I during the synthesis of fibril-forming collagen type I, has been associated with myocardial fibrosis. Myocardial fibrosis is a major determinant of both systolic and diastolic function of the heart. We hypothesize that differential degrees of myocardial fibrosis may be responsible for these discrepancies.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of left ventricular systolic dysfunction (measured LVEF% less than 35%) measured by echocardiography within the previous three months at the time of enrollment
2. Greater than or equal to 18 years of age
3. Greater than or equal to 110 pounds in weight

Exclusion Criteria:

1.Non-sinus rhythm at the time of enrollment

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Persons with left ventricular systolic dysfunction from the Texas Tech University Health Sciences Center outpatient clinic and University Medical Center, Lubbock, Texas
Sampling Method: Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
There will be a significant relationship between the severity of diastolic dysfunction and PICP

CONTACTS AND LOCATIONS:
Overall Officials: Chanwit Roongsritong, MD, Principal Investigator — TTUHSC
Locations (1):
- TTUHSC, Lubbock, Texas, United States